CLINICAL TRIAL: NCT02060578
Title: DELI-DEVI : Determinants of End-of-life Place of Care for Children Suffering From Cancer.
Brief Title: Determinants of End-of-life Place of Care for Children Suffering From Cancer.
Acronym: DELI-DEVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: University of Rennes 2 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 35RC13_9749_DELI-DEVI; 13.04.08 (Other: CPP Ouest III (Poitiers)); 13.428 (Other: CCTIRS); 913434 (Other: CNIL)
Record Dates: First submitted 2014-01-17; First posted 2014-02-12 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Cancer
Keywords: Cancer palliative care; Dead child
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Other): Questionnaire completed by the parents Interview with the parents and the psychologist (University Rennes 2)
  Interventions: Other: Questionnaire and interview

INTERVENTIONS:
Other: Questionnaire and interview — Questionnaire completed by the parents Interview with the parents and the psychologist (University Rennes 2)

SUMMARY:
Cancer is the second cause of over-one-year-old children mortality after accident. Survival rate is more than 70%, but in some cases, curative treatments are not sufficient and palliative support is implemented for those children in end of life.

Pediatric guidelines about the place of end-of-life care are varied. On European scale, home is recommended (IMPaCCT study, 2007). In France, the 2008-2012 palliative care development program recommended home or initial hospital care unit. This program also supports implementation of mobile team rather than specific hospital units.

In Brittany, a pattern of regional palliative care resource team has been implemented since 2005. In oncology, further to the guidelines, end-of-life place of care is often discussed several times for each case. Sometimes occur a lot of returns between home and hospital, psychological difficulties, and difficulties to offer adapted care conditions. Finally, less than 30% of children in palliative care decease at home.

The primary objective is to identify main determinants of the place of palliative care in pediatric oncology.

The secondary objective is to clarify the factors of change comparing to the initial planned place.

Intervention :

Questionnaire completed by the parents Interview with the parents and the psychologist (University Rennes 2)

Number of subjects is : Parents of 68 to 93 children who died from cancer after a palliative phase, that means 136 to 186 parents.

Expected results and perspectives :

Using both quantitative and qualitative methods, expected results are the followings:

* Identification of the objective and subjective factors, which influenced the decision of the place of care.
* Determination of the factors of change comparing to the initial planned place.

Once identified, main factors could be the ones to pay attention to in order to help for initial decision, better anticipation of change of place and better guidance of palliative care organization wherever, at home or in hospital.

Results would be new information for research on palliative care for children but also for adults.

Finally, this work is part of an improving approach of palliative care, related to the development of open-care hospital networks. We can expect some public health impacts with new arguments to help for complementary recommendations.

DETAILED DESCRIPTION:
Eligibility criteria :

Inclusion criteria are :

Parents of a deceased child

* From cancer, after palliative phase
* Age of death under 18 years old.
* Death occurred in Brittany
* Death between 2005 and 2010

Exclusion criterium is :

Parents of child who deceased after 2010 (respecting a bereavement delay)

Outcomes measures :

Primary study endpoint : Consideration or not by parents that they and/or their child had the choice of the end-of-life place of care.

Secondary study endpoints :

* objective factors : grade, occupational categories, marital status of parents, siblings, home conditions, access to the hospital, meeting with a professional of palliative care network, helpful general practitioner, volunteers, psychological support but also unexpected symptoms, needed nursing care which can explain a return from home to hospital for instance.
* subjective factors such as family or religious values, needs of intimacy, communication, support, sense of security, anxiety, fear, doubts about the next events.

ELIGIBILITY:
Inclusion Criteria:

Parents of a deceased child

* From cancer, after palliative phase
* Age of death under 18 years old.
* Death occurred in Brittany
* Death between 2005 and 2010

Exclusion Criteria:

Parents of child who deceased after 2010 (respecting a bereavement delay)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Consideration or not by parents that they and/or their child had the choice of the end-of-life place of care. | interview day
  Consideration or not by parents that they and/or their child had the choice of the end-of-life place of care.

SECONDARY OUTCOMES:
Objective factors | Interview day
  Objective factors : grade, occupational categories, marital status of parents, siblings, home conditions, access to the hospital, meeting with a professional of palliative care network, helpful general practitioner, volunteers, psychological support but also unexpected symptoms, needed nursing care which can explain a return from home to hospital for instance
Subjective factors | Interview day
  Subjective factors such as family or religious values, needs of intimacy, communication, support, sense of security, anxiety, fear, doubts about the next events.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Robert, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, Brittany Region, France